CLINICAL TRIAL: NCT01332552
Title: A Randomized, Double Blind, Dose Escalation, Fusion, First Time in Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Single and Repeat Doses of GSK2485852 in Chronically Infected Hepatitis C Subjects
Brief Title: A First Time in Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Single and Repeat Doses of GSK2485852 in Chronically Infected Hepatitis C Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to unfavorable human pharmacokinetic properties
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 115040
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C
Keywords: pharmacokinetics; First administration to human; antiviral activity; safety; hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — GSK2485852; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: Single dose escalation (Experimental): GSK2485852 planned single doses are placebo, 70 mg, 420 mg, 70 mg with food
  Interventions: Drug: GSK2485852 70 mg; Drug: GSK2485852 420 mg; Drug: placebo; Drug: GSK2485852 70 mg + Ritonavir 100mg
- Part 2: Repeat dose escalation (Experimental): GSK2485852 planned repeat doses are placebo, 420mg BID, 420mg TID, 630mg BID
  Interventions: Drug: placebo; Drug: GSK2485852 420 mg; Drug: GSK2485852 630 mg; Drug: GSK2485852 210 mg + Ritonavir 100mg
- Part 3: GSK2485852 + Ritonavir (Experimental): GSK2485852 single dose 70mg, 210 mg +Ritonavir 100mg x 1 day; GSK2485852 210mg + Ritonavir 100mg single dose x 3 days;
  Interventions: Drug: GSK2485852 210 mg +Ritonavir 100mg

INTERVENTIONS:
Drug: GSK2485852 70 mg — single dose
  Arms: Part 1: Single dose escalation
Drug: GSK2485852 420 mg — single dose
  Arms: Part 1: Single dose escalation
Drug: placebo — single dose
  Arms: Part 1: Single dose escalation
Drug: placebo — Repeat dose, once daily for 3 days
  Arms: Part 2: Repeat dose escalation
Drug: GSK2485852 420 mg — Repeat dose, twice daily for 3 days
  Arms: Part 2: Repeat dose escalation
Drug: GSK2485852 420 mg — Repeat dose, TIDfor 3 days
  Arms: Part 2: Repeat dose escalation
Drug: GSK2485852 630 mg — Repeat dose, twice daily for 3 days
  Arms: Part 2: Repeat dose escalation
Drug: GSK2485852 70 mg + Ritonavir 100mg — single dose, day 1
  Arms: Part 1: Single dose escalation
Drug: GSK2485852 210 mg + Ritonavir 100mg — single dose, day 1
  Arms: Part 2: Repeat dose escalation
Drug: GSK2485852 210 mg +Ritonavir 100mg — single dose daily for 3 days
  Arms: Part 3: GSK2485852 + Ritonavir

SUMMARY:
GSK2485852 is a Hepatitis C NS5B site IV non-nucleoside polymerase inhibitor being developed for the treatment of chronic HCV infection. HBI115040 is the first administration of GSK2485852 in humans to establish the initial safety, tolerability, pharmacokinetic, and antiviral profile. The study design is a fusion of single and repeat dosing cohorts in HCV infected subjects to evaluate the safety, pharmacokinetics, and antiviral activity of GSK2485852.

HBI115040 describes a Phase I, randomized, double-blind, placebo-controlled, dose escalation fusion study to determine the safety, tolerability, pharmacokinetic, and antiviral profile of GSK2485852 in single doses (Part 1), repeat doses (Part 2), and ritonavir co-administration (Part 3) in chronically infected HCV subjects. The study will also explore the effect of a moderate (30%) fat meal on pharmacokinetic endpoints in HCV subjects in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply: Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring (i.e., ECG), including no cardiac, pulmonary, hepatic, biliary, gastrointestinal, or renal disorders, or cancer within the past 5 years.
* Males or females between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential.
* Body weight > or = 50 kg (110 lbs.) for men and > or = 45 kg (99 lbs.) for women and BMI between 18.5-35.0 kg/m2 inclusive will be allowed.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* AST, ALT, and alkaline phosphatase <3.0xULN and bilirubin <1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Average QTcB or QTcF < 450 msec; or QTcB or QTcF < 480 msec in subjects with Bundle Branch Block.
* Treatment naive chronically infected HCV subjects, defined as infection for >6 months and no prior HCV therapy, with an HCV RNA viral load of greater than 100,000 IU/mL and HCV genotype 1a or 1b. HCV subjects with mixed genotypes are not eligible for the study.
* Positive for HCV RNA and anti-HCV antibody at the time of screening AND positive for anti-HCV antibody, HCV RNA, or an HCV genotype at least 6 months before screening; OR Positive for HCV RNA and anti-HCV antibody at the time of screening AND liver biopsy within three years prior to screening indicating the absence of cirrhosis.

Exclusion Criteria:

* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* A positive pre-study Hepatitis B surface antigen or HIV antibody within 3 months of screening.
* A positive pre-study drug/alcohol screen.
* History of regular alcohol consumption within 6 months of the study.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer). Exposure to more than four new investigational products within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication,
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Holter monitoring shows one or more of the following: Any symptomatic arrhythmia (except isolated extra systoles); Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, SVT (>10 consecutive beats)); Sustained tachycardia >150 beats per minute; Non-sustained or sustained ventricular tachycardia (defined as >3 consecutive ventricular ectopic beats); Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher in an awake subject], WPW syndrome, other pre-excitation syndromes); Symptomatic sinus pause or sinus pause >3 seconds - unless patient is straining, vomiting, or having some other type of hypervagal response; 300 or more supraventricular ectopic beats in 24 hours; 250 or more ventricular ectopic beats in 24 hours; Ischemia, diagnosed by a sequence of ECG changes that include flat or downsloping ST-segment depression >0.1 mV, with a gradual onset and offset that lasts for a minimum period of 1 minute. Each episode of ischemia must be separated by a minimum duration of at least 1 minute, during which the ST segment returns back to baseline (1x1x1 rule).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-01-14 (Actual); Primary Completion 2011-04-06 (Actual); Study Completion 2011-04-06 (Actual)

PRIMARY OUTCOMES:
Safety parameters: adverse events; telemetry; absolute values and changes over time of hematology, clinical chemistry, urinalysis, vital signs (blood pressure, heart rate), and electrocardiogram (ECG) parameters | up to 7 days
GSK2485852 PK parameters following single dose administration: AUC(0-inf), AUC(0-t), AUC(0-24), Cmax, tmax, C24, t1/2, tlag, and CL/F | 24 hours
GSK2485852 PK parameters following repeat dose administration: AUC(0-τ), Cτ, Cmax, tmax, t1/2, and CL/F | 72 hours
HCV RNA viral load reduction from baseline | 24 to 72 h
HCV RNA change from baseline to nadir | up to 72 h
Time course of HCV viral load at baseline, during dosing with GSK2485852, and > or = 14 days after GSK2485852 dosing | up to 14 days

SECONDARY OUTCOMES:
GSK2485852 PK parameters: AUC(0-24), Cmax, tmax and tlag following a single dose with and without moderate fat/calorie meal. | 24 h
GSK2485852 accumulation ratio (R) | 72 h
GSK2485852 time invariance in non-food cohorts | 72 hours
GSK2485852 dose proportionality after single or repeat dosing in non-food cohorts | up to 72 h

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Willingboro, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115040 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115040?search=study&search_terms=115040#rs
- Available data/document: Informed Consent Form: 115040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register